CLINICAL TRIAL: NCT07391553
Title: What Are the Isokinetic Strength Outcomes and Self-reported Functional Outcomes (ATRS) at 12 Months Following Non-surgical Management of Achilles Tendon Rupture Using the SMART Protocol?
Brief Title: Achilles Tendon Rupture Patient Outcomes at 12 Months
Acronym: ATR-12
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Raymond Healy, Senior Physiotherapist, Liverpool University Hospitals NHS Foundation Trust
Other Study IDs: JRO-0663; IRAS ID: 357432 (Other: Health Research Authority); JRO-0663 (Other: LIVERPOOL HEALTH PARTNERS JOINT RESEARCH OFFICE)
Record Dates: First submitted 2026-01-25; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture; Physiotherapy; orthopaedics; trauma; rehabilitation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Surgically Managed Achilles Tendon Rupture Cohort: Adults who sustained an Achilles tendon rupture and were managed non-surgically using the SMART rehabilitation protocol within Liverpool University Hospitals NHS Foundation Trust. All participants are 12-15 months post-injury at the time of assessment.
  Interventions: Other: Non-Surgical Management Using the SMART Protocol

INTERVENTIONS:
Other: Non-Surgical Management Using the SMART Protocol — Participants previously received standard non-surgical treatment for Achilles tendon rupture following the SMART (Swansea Morriston Achilles Rupture Treatment) functional rehabilitation protocol as part of routine NHS care. No interventions are assigned as part of this study; all data are collected at a single follow-up visit.

SUMMARY:
The Achilles tendon is the strongest and largest tendon in the human body, playing a critical role in plantarflexion and facilitating activities such as walking, running, and jumping. However, it is also the most frequently ruptured tendon. The injury and associated disability have a significant impact on patient quality of life and healthcare services. Achilles tendon ruptures are increasingly common, particularly among middle-aged recreational athletes, with an incidence estimated at 18 per 100,000 person-years.

The Swansea Morriston Achilles Rupture Treatment (SMART) protocol represents a structured, progressive approach to non-operative rehabilitation. It emphasizes early mobilization, protected weight-bearing, and a gradual return to sport or high-level function through targeted strength and neuromuscular training. While short-term outcomes of non-surgical protocols have demonstrated promising results, there remains limited high-quality data on long-term isokinetic strength and patient-reported functional outcomes beyond six months in this patient group.

This study aims to evaluate isokinetic plantarflexor strength and self-reported functional outcomes at 12 months following non-surgical management of Achilles tendon ruptures using the SMART rehabilitation protocol. By assessing both objective and subjective recovery metrics, we aim to contribute to the growing evidence base for evidence-informed, conservative Achilles tendon rehabilitation. A secondary aim of the study is to examine the relationship between isokinetic strength scores and self reported functional recovery scores using the ATRS questionnaire.

Participants will attend one 60-90 minute visit to complete a short questionnaire and perform a safe, clinic-based ankle strength test using an isokinetic machine; the test feels like pushing against a footplate, similar to resisted ankle movements. The results of these tests will be collected and analysed. The study will help to gain further insight into patient recovery from this injury.

DETAILED DESCRIPTION:
Background and Rationale Achilles tendon rupture (ATR) is a common injury in active adults and is increasingly managed non-surgically using structured, functional rehabilitation pathways. The Swansea Morriston Achilles Rupture Treatment (SMART) protocol is a widely implemented conservative pathway emphasising protected weight-bearing, staged mobilisation, and progressive strengthening. Although early functional outcomes with non-surgical care are encouraging, there remains limited single-time-point data at ~12 months post-injury combining objective plantarflexor strength with patient-reported function in routine NHS practice. This cross-sectional observational study addresses that gap by quantifying isokinetic strength and self-reported outcomes at 12-15 months after ATR managed non-operatively.

Objectives Primary objectives are to (1) quantify plantarflexor strength of the injured limb (peak torque and peak torque normalised to bodyweight) and (2) estimate recovery using Limb Symmetry Index (LSI) relative to the contralateral limb; and (3) describe patient-reported function using the Achilles Tendon Total Rupture Score (ATRS). A secondary objective is to examine the association between objective strength metrics and ATRS.

Design and Setting This is a single-organisation, cross-sectional cohort study conducted within Liverpool University Hospitals NHS Foundation Trust (LUHFT), with testing delivered at Aintree University Hospital or Broadgreen Hospital physiotherapy departments. Each participant attends one study visit (approximately 60-90 minutes). No randomisation, blinding, investigational product, or longitudinal follow-up is involved.

Study Population and Identification Adults (≥18 years) with a confirmed ATR treated non-surgically using the SMART protocol and now 12-15 months post-injury are identified by authorised clinicians from an existing LUHFT clinical database. Potential participants are approached by their direct care team or via text and provided with a Letter of Invitation and Participant Information Leaflet. Written informed consent is obtained prior to any study procedures.

Study Procedures Pre-test instructions: Participants are asked to avoid vigorous lower-limb activity for 24 hours pre-visit.

Warm-up: ~5 minutes of gentle cycling at a self-selected pace to elevate heart and breathing rate while maintaining conversational effort.

Isokinetic Strength Testing: Conducted with a clinic isokinetic dynamometer in a semi-reclined position with knee flexed to ~90°. The ankle joint is aligned with the dynamometer axis; the foot is strapped to the footplate; trunk/pelvis/thigh stabilised with padded straps. Testing range spans approximately 15° dorsiflexion to 40° plantarflexion. After sub-maximal familiarisation repetitions, participants perform maximal-effort concentric plantarflexion contractions at 90°/s and 30°/s on the uninjured limb first, then the injured limb.

Patient-Reported Outcome: Participants complete the ATRS (0-100; higher scores indicate better function).

Risk Management and Safety Monitoring The procedures are low-risk and part of routine rehabilitation assessment. Minor, transient muscle soreness (DOMS) or fatigue may occur. Testing is supervised by trained physiotherapists and is stopped immediately if pain or undue discomfort is reported. Any adverse events during the visit are documented and handled per local clinical governance; related and unexpected serious events would be reported to the sponsor and REC in line with policy.

Data Elements and Outcomes:

Objective outcomes include peak plantarflexion torque (Nm), peak torque normalised to bodyweight (Nm/kg), and LSI (%) calculated as (injured/uninjured) × 100. Subjective outcome is ATRS (0-100). Data are collected at a single time point only (12-15 months post-injury).

Sample Size and Feasibility A paired comparison of injured vs. uninjured limbs informed the sample size. Assuming 80% power (α=0.05), 92 participants were required to detect a clinically meaningful difference in peak torque; to allow for unusable data or non-completion, the target enrolment is 115.

Sampling Method Convenience sampling from the pre-existing clinical database of eligible ATR patients managed non-surgically with SMART in LUHFT. This approach reflects real-world NHS practice and facilitates operational feasibility for a single-visit assessment.

Statistical Analysis Plan Descriptive statistics will summarise all outcomes. Normality will be assessed. Between-limb comparisons for peak torque may be summarised descriptively; LSI will be presented as percentage. Association between strength metrics (peak torque, Nm/kg, and LSI) and ATRS will be assessed with Pearson's correlation when assumptions are met; otherwise, Spearman's rank correlation will be used. No imputation is planned; missing data will be described and analyses conducted on available data. All analyses are exploratory and hypothesis-generating within a cross-sectional framework.

Data Quality and Management Data are recorded on standardised case report forms and transferred to a secure, password-protected NHS server. Identifiable information is stored separately from research data; a study ID links records. Data entry checks and plausibility rules (e.g., range checks for torque values, internal consistency across speeds and limbs) are applied. Source documentation (e.g., printouts from the isokinetic system) is retained in site files. Only authorised staff have access to identifiable data. Pseudonymised datasets are used for analysis. No data are transferred outside approved secure environments.

Confidentiality and Governance The study complies with UK GDPR and the Data Protection Act 2018. Participation is voluntary and withdrawal can occur at any time without impact on care. Publications and presentations will report only aggregated, anonymised results; no individual-level data will be publicly shared.

Dissemination:

Findings will be submitted to peer-reviewed journals and presented at relevant conferences. Participants may opt to receive a lay summary of study results after analysis is complete.

Current Status:

Single-visit assessments will commence after all approvals and registrations are in place. Recruitment will continue until the planned sample size is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at the time of recruitment.
* Confirmed diagnosis of Achilles tendon rupture, diagnosed clinically and recorded within the NHS database.
* Injury managed non-surgically using the SMART (Swansea Morriston Achilles Rupture Treatment) protocol.
* 12-15 months post-injury at the time of assessment.
* Able and willing to provide informed written consent to participate in the study.

Exclusion Criteria:

* Unable to provide informed consent.
* Previous surgical repair of the Achilles tendon or documented re-rupture.
* Presence of a neuromuscular disorder affecting lower limb strength or function.
* Did not follow the SMART protocol for non-surgical management.
* History of Achilles tendinopathy or rupture in the contralateral (uninjured) leg.
* Unable to tolerate isokinetic strength testing due to pain, discomfort, or other medical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who previously sustained an Achilles tendon rupture and were treated non-surgically using the SMART rehabilitation protocol within Liverpool University Hospitals NHS Foundation Trust. Eligible participants are identified from an existing clinical database and represent patients 12-15 months post-injury who completed standard physiotherapy rehabilitation. All participants are drawn from routine NHS orthopaedic and physiotherapy services at Aintree and Broadgreen Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Peak Plantarflexion Torque (Nm) | 12-15 months post-injury (single study visit)
  Maximum rotational force produced by the plantarflexor muscles during an isokinetic concentric contraction, measured using an isokinetic dynamometer. This measure reflects calf muscle strength and tendon function following non-surgical Achilles tendon rupture management.
Peak Plantarflexion Torque Normalized to Bodyweight (Nm/kg) | 12-15 months post-injury (single study visit)
  Peak plantarflexion torque adjusted for each participant's bodyweight. Normalisation allows strength comparisons between individuals of different body sizes and provides a more functional evaluation of recovery.
Limb Symmetry Index (LSI) for Peak Torque (%) | 12-15 months post-injury (single study visit)
  Ratio of injured limb peak plantarflexion torque to the uninjured limb, expressed as a percentage. An LSI ≥90% is typically considered indicative of satisfactory recovery.
Achilles Tendon Total Rupture Score | 12-15 months post-injury (single study visit)
  A validated patient-reported outcome measure assessing symptoms and functional limitations following Achilles tendon rupture. Scores range from 0 to 100, with higher scores indicating better perceived recovery.

SECONDARY OUTCOMES:
Correlation Between Isokinetic Strength Measures and Achilles Tendon Total Rupture Score | 12-15 months post-injury (single study visit)
  Statistical correlation between objective isokinetic strength metrics (peak torque, PT:BW, and LSI) and subjective functional recovery measured by ATRS. Pearson's correlation coefficient will be used unless data violate normality assumptions, in which case Spearman's rank correlation will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Morton, BSc. (Hons) Physiotherapy, Study Chair — Liverpool University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Broadgreen Hospital Physiotherapy department, Liverpool, Merseyside
  - Aintree University Hospital Therapies department, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregated, anonymised results will be published. This is consistent with participant consent and NHS data governance requirements

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol with NCT number (2026-02-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT07391553/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol prior to PRS review (2026-01-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT07391553/Prot_SAP_000.pdf
  • Informed Consent Form (2026-01-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT07391553/ICF_001.pdf